CLINICAL TRIAL: NCT06077422
Title: Randomized Control Trial to Assess the Efficacy of Preoperative Erector Spinae Blocks on Cardiac Surgery Postoperative Outcomes
Brief Title: Exparel vs. Marcaine ESP Block for Post-cardiac Surgical Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Leonard Y. Lee, MD, James W. Mackenzie, M.D. Professor and Chair, Department of Surgery, Rutgers Robert Wood Johnson Medical School, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2022001580
Record Dates: First submitted 2023-07-15; First posted 2023-10-11 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative; Opioid Use; Perioperative Complication; Heart Diseases
Keywords: plane block; sternotomy; thoracotomy; cardiac; surgery; postoperative; pain; anesthesia; opioid; pragmatic trial
MeSH Terms: conditions — Pain, Postoperative; Heart Diseases; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exparel (Experimental): The experimental medication (Exparel) will be administered per standard of care via ultrasound-guided erector spinae plane (ESP) blocks, bilaterally for sternotomy and unilaterally for mini-thoracotomy. The drug will be administered prior to cardiac surgery. The dosage will be determined by patient body weight.
  For this pilot project the investigators anticipate consenting 120 subjects to obtain 96 evaluable subjects; 48 Mini thoractomies (N=24 Exparel, N=24 Marcaine) 48 Open sternotomies (N=24 Exparel, N=24 Marcaine).
  Interventions: Drug: bupivacaine liposome injectable suspension
- Marcaine (Active Comparator): The active comparator medication (Marcaine) will be administered per standard of care via ultrasound-guided erector spinae plane (ESP) blocks, bilaterally for sternotomy and unilaterally for mini-thoracotomy. The drug will be administered prior to cardiac surgery. The dosage will be determined by patient body weight.
  For this pilot project the investigators anticipate consenting 120 subjects to obtain 96 evaluable subjects; 48 Mini thoracotomies (N=24 Exparel, N=24 Marcaine) 48 Open sternotomies (N=24 Exparel, N=24 Marcaine).
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: bupivacaine liposome injectable suspension — Bupivacaine liposome injectable suspension (Exparel) will be administered by ultrasound-guided ESP block, unilaterally if thoracotomy on ipsilateral side, bilaterally if median sternotomy.
  Other Names: Exparel
  Arms: Exparel
Drug: Bupivacaine Hydrochloride — Bupivacaine HCl (Marcaine) will be administered by ultrasound-guided ESP block, unilaterally if thoracotomy on ipsilateral side, bilaterally if median sternotomy.
  Other Names: Marcaine
  Arms: Marcaine

SUMMARY:
The goal of this pilot study is to describe and compare Ultrasound-Guided Erector Spinae Plane (ESP) Blocks using Exparel® (bupivacaine liposome injectable suspension) to Marcaine® (bupivacaine hydrochloride) for pain management and outcomes after cardiac surgeries.

DETAILED DESCRIPTION:
Postoperative pain is a major concern for patients after cardiovascular surgery.

With an increasing emphasis on improving perioperative care arising from evidence-based protocols such as Enhanced Recovery After Surgery (ERAS), reducing postoperative pain not only increases patient satisfaction, but also decreases postoperative complications and improves outcomes. Reduced postoperative pain also decreases rates of pneumonia and time on mechanical ventilation, in the ICU, or in the hospital. Importantly, decreasing postoperative pain can also reduce high dose opioid usage, the established method of managing postoperative pain, thereby decreasing rates of nausea/vomiting, intubation time, and mortality. Methods of reducing postoperative pain, such as neuraxial anesthesia and deep plexus blocks, are associated with an increased risk of epidural hematoma; an alternate solution, therefore, is using fascial plane blocks.

Since 2018, our institution is one of very few that uses pre-operative fascial plane blocks for cardiac surgery patients, implementing bilateral plane blocks for the sternotomy approach and unilateral plane blocks for the right mini-thoracotomy approach. Results from these blocks have been quite favorable but not yet validated.

A study in which subjects are randomized to not receive an ESP block preoperatively would raise concerns regarding equipoise. Therefore, this study is designed to better understand the overall effects of these blocks by comparing FDA approved medications, Exparel (current practice at RWJUH) and Marcaine. Marcaine (0.25% bupivacaine HCl) has an onset of action on the order of seconds and generally within one minute from the time of injection, and an effect duration of roughly seven hours. Exparel is a commercially available extended-release formulation of liposomal bupivacaine, which extends the effect duration to an upward of 72 hours from the time of injection with similarly immediate onset of action. Several studies have compared local injections of Marcaine (plain bupivacaine) with Exparel (liposomal bupivacaine) in the setting of inguinal hernia repair, knee arthroplasty, breast augmentation, and hemorrhoidectomy, with results favoring the use of liposomal bupivacaine based on improvements in subjective pain at the initial postoperative pain assessment.(6) Clinical trials are currently underway, investigating the effect of liposomal bupivacaine for local anesthesia and compared with epidural anesthesia in thoracoscopic surgery. In a recent clinical trial published in the Journal of the American Medical Association (JAMA), patients undergoing cardiothoracic or vascular surgery subjected to truncal incisions did not demonstrate a significant benefit with respect to pain control or adjunctive opioid usage when treated with liposomal bupivacaine over plain bupivacaine via local injection. Still, a gap in the literature exists with respect to the use of liposomal bupivacaine versus plain bupivacaine for erector spinae plane block in the setting of sternotomy. The aim of this prospective study is to determine the impact of preoperative fascial plane blocks with Exparel compared to Marcaine on outcomes following cardiac procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years-no upper age limit)
* Scheduled for mini thoracotomy (i.e. valve repair) or open sternotomy (i.e. bypass graft) at single academic medical center (in and out-patients).

Exclusion Criteria:

Patients will be excluded if they:

* Are currently on pain medication or pain regimen for chronic pain condition
* Convert to sternotomy (for thoracotomies)
* Require, upon intraoperative discovery and surgeon's decision, the need for an unplanned secondary procedure other than the originally scheduled index operation
* Undergo emergent surgery
* Are non-English speaking (The majority of the PI's patient population speak English. As a pilot study the investigators cannot afford to enroll non-English speaking subjects due to time, personnel, and financial constraints.)
* Mechanical circulatory support (MCS)
* Vasoactive medications
* Intubated
* Active infection
* Patients otherwise deemed ineligible for ESP block by the investigators due to safety concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Postoperative days 0 through 5
  Postoperative opioid consumption within first five postoperative days, reported as average mg/day in morphine equivalents.

SECONDARY OUTCOMES:
Postoperative nonopioid analgesic consumption | Postoperative days 0 through 5
  Postoperative non-opioid analgesic (Pregabalin, Gabapentin, selective serotonin reuptake inhibitor (SSRI), selective norepinephrine reuptake inhibitor (SNRI), Ketorolac, Tramadol, Ibuprofen, and Acetaminophen) consumption within first five postoperative days, reported as average mg/day.
Inpatient postoperative pain score | Postoperative days 0 through 5
  Pain scores through postoperative day five, using the standard Numeric Rating Scale (NRS), wherein a score of 0 corresponds to "no pain," 5 to "moderate pain," and 10 to "worst possible pain," reported as mean score over all five days.
Outpatient postoperative pain score | Obtained within 30 days following surgery
  Single pain score at follow-up visit, using the standard Numeric Rating Scale (NRS), wherein a score of 0 corresponds to "no pain," 5 to "moderate pain," and 10 to "worst possible pain."
30-day mortality rate | Through postoperative day 30
  Proportion of patients who expire within 30 postoperative days from the index operation.
30-day major morbidity rate | Through postoperative day 30
  Proportion of patients who experience the composite outcome of major morbidity, defined as the occurrence of any of the following within 30 postoperative days from the index operation: pneumonia, respiratory failure with ventilatory support >48h, pulmonary embolism (PE), deep vein thrombosis (DVT), multi-organ dysfunction syndrome, postoperative myocardial infarction (MI), acute renal failure requiring renal replacement therapy, cerebrovascular accident (CVA), infection of wound or line or urinary tract infection (UTI), readmission, sustained postoperative atrial or ventricular arrhythmia, new postoperative atrial fibrillation, exacerbation of pre-existing atrial fibrillation
Postoperative qualify of life | Within the range of 30 days prior to surgery to 30 days after surgery
  Measured as change on the 12-item Short Form Survey (SF-12) from preoperative baseline to followup. Scores on the SF-12 range from 0 to 100, with higher scores indicating better physical and mental health.
Hospitalization cost | Study duration, limited to one year.
  Before-insurance cost of hospitalization and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Y Lee, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School, Dept of Surgery
Locations (1):
- Rutgers RWJMS, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toscano A, Barbero C, Capuano P, Costamagna A, Pocar M, Trompeo A, Pasero D, Rinaldi M, Brazzi L. Chronic postsurgical pain and quality of life after right minithoracotomy mitral valve operations. J Card Surg. 2022 Jun;37(6):1585-1590. doi: 10.1111/jocs.16400. Epub 2022 Mar 11. PMID 35274774
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Background] Song K, Xu Q, Knott VH, Zhao CB, Clifford SP, Kong M, Slaughter MS, Huang Y, Huang J. Liposomal Bupivacaine-Based Erector Spinae Block for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 May;35(5):1555-1559. doi: 10.1053/j.jvca.2020.09.115. Epub 2020 Sep 20. No abstract available. PMID 33046362
- [Background] Collins JB, Song J, Mahabir RC. Onset and duration of intradermal mixtures of bupivacaine and lidocaine with epinephrine. Can J Plast Surg. 2013 Spring;21(1):51-3. doi: 10.1177/229255031302100112. PMID 24431939
- [Background] Gadsden J, Long WJ. Time to Analgesia Onset and Pharmacokinetics After Separate and Combined Administration of Liposome Bupivacaine and Bupivacaine HCl: Considerations for Clinicians. Open Orthop J. 2016 Apr 12;10:94-104. doi: 10.2174/1874325001610010094. eCollection 2016. PMID 27347237
- [Background] Sandhu HK, Miller CC 3rd, Tanaka A, Estrera AL, Charlton-Ouw KM. Effectiveness of Standard Local Anesthetic Bupivacaine and Liposomal Bupivacaine for Postoperative Pain Control in Patients Undergoing Truncal Incisions: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e210753. doi: 10.1001/jamanetworkopen.2021.0753. PMID 33724391
- See also: Exparel and Marcaine for Pain Management in Thoracoscopic Lobectomy Patients (BEMP) — https://classic.clinicaltrials.gov/ct2/show/NCT03682224
- See also: Study of Exparel Versus Epidural for Pain Control After Thoracotomy — https://clinicaltrials.gov/ct2/show/NCT02178553

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT06077422/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT06077422/ICF_003.pdf